CLINICAL TRIAL: NCT06282081
Title: Serum Neurofilament Light As a Clinical Tool in Relapsing Remitting Multiple Sclerosis
Brief Title: Serum Neurofilament Light in Multiple Sclerosis
Status: Active, not recruiting | Type: Observational
Sponsor: Dent Neuroscience Research Center (Other)
Collaborators: Genentech, Inc., a subsidiary of F. Hoffman-La Roche AG (Unknown); Monogram Biosciences (LabCorp Specialty Testing Group) (Unknown)
Responsible Party: Sponsor
Other Study IDs: ML 45098
Record Dates: First submitted 2024-02-02; First posted 2024-02-28 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis; Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Serum Neurofilament Light — The purpose of this research is to investigate a biomarker, called serum neurofilament light (sNfL), which is measured in blood. This study will attempt to investigate whether or not sNfL is a useful tool for clinicians in patients diagnosed with relapsing remitting multiple sclerosis.

SUMMARY:
This prospective cohort study is designed to characterize the utility of sNfL as a biomarker in clinical practice. This study also aims to understand how access to sNfL measures affects patient and clinician knowledge of their disease status and capture how this may have the potential to influence clinical decision-making. Level of disability, cognitive changes, fatigue, depression, and quality of life to detect clinical and subclinical worsening will be measured. While there is strong evidence in support of sNfL as a potential biomarker, literature regarding the application of sNfL in a real-world clinical practice setting is lacking. Understanding the utility of this test to clinicians and patients as a biomarker of MS disease activity is essential. Additionally, the optimum sampling frequency in clinical practice should be investigated to further elucidate its practicality. Given recent advances in the treatment of MS, there is increasing need for convenient and accessible measures of treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with RRMS
2. Adults aged 18+ at time of screening
3. Patients who are able to consent
4. Patients who agree to be reasonably compliant with study protocol for the duration of the study
5. Any subject who is currently being treated with an MS DMT or any subject initiating a new MS DMT throughout the duration of their participation in the study will be initiated and/or treated according to local label

Exclusion Criteria:

1. Patients with current diagnosis of a neurodegenerative or autoimmune disease other than MS that may impact sNfL levels, in the opinion of the investigator (including but not limited to: Alzheimer's disease, Huntington's disease, Amyotrophic Lateral Sclerosis, or Parkinson's disease, systemic lupus erythematosus, rheumatoid arthritis)
2. Inability to complete blood draws
3. Pregnant or breastfeeding, or planning to become pregnant or breastfeed for the duration of the study
4. Patients who have taken an investigational medication within five half-lives prior to screening or who plan to take an investigational medication during the study
5. Patients with a medical condition or taking a medication that may interfere with study endpoints in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with relapsing remitting multiple sclerosis.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the utility of sNfL levels to aid with clinical decision-making by examining clinicians' understanding of patient's clinical status before sNfL results are received vs. after sNfL results are received | 1 year
  This outcome is based on structured clinician questionnaires developed for this study. Prior to receiving patient sNfL results, clinicians will answer the question "My current clinical impression of this patient's disease status is (circle one): a. Stable, b. Suspected disease activity, c. Confirmed disease activity, d. At risk for relapse, e. Relapse, f. Other (please specify)." After receiving patient sNfL results, clinicians will answer the question "After reviewing this patient's sNfL results along with other diagnostic testing at this time, my opinion of the patient's disease status is (circle one): a. Stable, b. Suspected disease activity, c. Confirmed disease activity, d. At risk for relapse, e. Relapse, f. Other (please specify)" and these answers will be reported.
Evaluate the utility of sNfL levels to aid with clinical decision-making by examining clinicians' opinion as to how sNfL results could guide clinical practice | 1 year
  This outcome is based on a structured clinician questionnaire developed for this study. Clinicians will answer the question: "This patient's sNfL results have had the following impact on my opinions or confidence in this patient's care plan, or have potential to guide my clinical practice in the following way (please list specifics, e.g., increased confidence in assessment of disease status; decision to order additional testing; change in mediation therapy; change in frequency of follow-up, etc)" and these answers will be reported.
Describe the optimal sNfL sampling frequency by capturing frequency of unscheduled clinician-ordered sNfL measurements. | 1 year
Describe the optimal sNfL sampling frequency by capturing reason for unscheduled clinician-ordered sNfL measurements. | 1 year
  This outcome is based on a structured clinician questionnaire developed for this study. Prior to receiving patient's sNfL results, clinicians will answer the question, "Is this an unscheduled sNfL measurement? Yes No; If yes, please specify reason why this sNfL measurement was scheduled" and these answers will be reported.
Describe the optimal sNfL sampling frequency by capturing usefulness of scheduled and unscheduled sNfL measurements based on a visual analog scale. | 1 year
  After receiving sNfL results, clinicians will answer the following prompt on a visual analog scale: "Knowledge of sNfL level has the potential to be useful in my clinical practice for this patient" and these answers will be reported. The scale is measured from "Not at all" to "extremely."
Describe the optimal sNfL sampling frequency by capturing usefulness of scheduled and unscheduled sNfL measurements based on a visual analog scale. | 1 year
  After receiving sNfL results, clinicians will answer the following prompt on a visual analog scale: "sNfL results has the potential to be a useful/suitable alternative to MRI for this patient" and these answers will be reported. The scale is measured from "Not at all" to "extremely."

SECONDARY OUTCOMES:
Describe patient demographics | 1 year
Describe patient comorbidities | 1 year
Describe patient concomitant medications | 1 year
Describe patient MS medications | 1 year
Describe patient reasons for MS medication changes | 1 year
Describe patient MS relapses including date of relapse | 1 year
Describe patient MS relapses including clinical findings | 1 year
Describe patient MS relapses including radiologic findings | 1 year
Describe patient MS relapses including severity | 1 year
  Severity of MS relapses will be described by change in EDSS score from non-relapsing EDSS measurement.
Explore patient attitudes towards sNfL measurements by capturing patients' perceptions of undergoing sNfL measurements vs. receiving an MRI based on a structured questionnaire. | 1 year
  This outcome is based on a structured patient questionnaire developed for this study. Patients will answer the following question after receiving sNfL results: "How much do you agree with the following statements on a scale of 0 to 10, where 0 is "completely disagree" and 10 is "completely agree"? Compared to MRI, sNfL draws were more accessible: ____________ " and these answers will be reported.
Explore patient attitudes towards sNfL measurements by capturing patients' perceptions of undergoing sNfL measurements vs. receiving an MRI based on a structured questionnaire. | 1 year
  This outcome is based on a structured patient questionnaire developed for this study. Patients will answer the following question after receiving sNfL results: "How much do you agree with the following statements on a scale of 0 to 10, where 0 is "completely disagree" and 10 is "completely agree"? Compared to MRI, sNfL draws were more burdensome: ___________" and these answers will be reported.
Explore patient attitudes towards sNfL measurements by capturing patients' perceptions of undergoing sNfL measurements vs. receiving an MRI based on a structured questionnaire. | 1 year
  This outcome is based on a structured patient questionnaire developed for this study. Patients will answer the following question after receiving sNfL results: "How much do you agree with the following statements on a scale of 0 to 10, where 0 is "completely disagree" and 10 is "completely agree"? Compared to MRI, sNfL draws were more uncomfortable: ___________" and these answers will be reported.
Explore patient attitudes towards sNfL measurements by capturing patients' perceptions of undergoing sNfL measurements vs. receiving an MRI based on a structured questionnaire. | 1 year
  This outcome is based on a structured patient questionnaire developed for this study. Patients will answer the following question after receiving sNfL results: "How much do you agree with the following statements on a scale of 0 to 10, where 0 is "completely disagree" and 10 is "completely agree"? Compared to MRI, sNfL draws were easier to fit into my schedule: ____________" and these answers will be reported.
Explore patient attitudes towards sNfL measurements by capturing patients' perceptions of undergoing sNfL measurements vs. receiving an MRI based on a structured questionnaire. | 1 year
  This outcome is based on a structured patient questionnaire developed for this study. Patients will answer the following question after receiving sNfL results: "How much do you agree with the following statements on a scale of 0 to 10, where 0 is "completely disagree" and 10 is "completely agree"? Compared to MRI, sNfL results were more difficult to understand: ____________" and these answers will be reported.
Explore patient attitudes towards sNfL measurements by capturing patients' understanding of their disease before sNfL results are received vs. after sNfL results are received via a structured questionnaire. | 1 year
  This outcome is based on structured patient questionnaires developed for this study. Patients will answer the following question before and after receiving sNfL results: "My current understanding of my MS disease is that I am (circle one): a. Stable, b. Experiencing increased disease activity, c. At risk for relapse, d. Experiencing a relapse, e. Unknown" and these answers will be reported.
Explore patient attitudes towards sNfL measurements by capturing patient attitudes towards sNfL sampling via a structured questionnaire. | 1 year
  This outcome is based on a structured patient questionnaire developed for this study. Patients will answer the following question after receiving sNfL results: "How much do you agree with the following statements on a scale of 0 to 10, where 0 is "completely disagree" and 10 is "completely agree"? sNfL results were easy to understand: _______" and these results will be reported.
Explore patient attitudes towards sNfL measurements by capturing patient attitudes towards sNfL sampling via a structured questionnaire. | 1 year
  This outcome is based on a structured patient questionnaire developed for this study. Patients will answer the following question after receiving sNfL results: "How much do you agree with the following statements on a scale of 0 to 10, where 0 is "completely disagree" and 10 is "completely agree"? sNfL results increased my knowledge of my MS disease status: ____________" and these results will be reported.
Compare sNfL levels after initiation of a new MS disease-modifying therapy (DMT; when patient is treated with a DMT) vs. prior to MS DMT initiation (when patient is not treated with any DMT) where available. | 1 year
Compare sNfL levels at scheduled sampling time points between patients initiating any new MS DMT vs. patients who do not change MS DMT where available. | 1 year
Compare sNfL levels in patients who have a clinical or radiologic relapse during the study vs. patients who do not. | 1 year
Describe changes in sNfL levels with Expanded Disability Status Scale (EDSS) where available. | 1 year
  EDSS scale is from 0 to 10, where 0 indicates normal neurologic exam and 10 indicates death due to MS.
Describe changes in sNfL levels with Symbol Digit Modalities Test (SDMT) where available. | 1 year
  SDMT scale is from 0 to 110, where 0 indicates none correct and 110 indicates all correct.
Describe changes in sNfL levels with Patient Health Questionnaire-9 (PHQ-9) where available. | 1 year
  PHQ-9 scores from 0 to 27, where 1-4 indicates minimal depression and 20-27 indicates severe depression.
Describe changes in sNfL levels with Multiple Sclerosis Quality of Life - 54 (MSQOL-54) physical health summary score where available. | 1 year
  MSQOL-54 scale scores range from 0 to 100 and a higher scale score indicates improved quality of life.
Describe changes in sNfL levels with Multiple Sclerosis Quality of Life - 54 (MSQOL-54) mental health summary score where available. | 1 year
  MSQOL-54 scale scores range from 0 to 100 and a higher scale score indicates improved quality of life.
Describe changes in sNfL levels with magnetic resonance imaging disease activity where available. | 1 year
Describe changes in sNfL levels with changes to multiple sclerosis disease-modifying therapy where available. | 1 year
Compare changes in sNfL levels with Expanded Disability Status Scale (EDSS) where available. | 1 year
  EDSS scale is from 0 to 10, where 0 indicates normal neurologic exam and 10 indicates death due to MS.
Compare changes in sNfL levels with Symbol Digit Modalities Test (SDMT) where available. | 1 year
  SDMT scale is from 0 to 110, where 0 indicates none correct and 110 indicates all correct.
Compare changes in sNfL levels with Patient Health Questionnaire-9 (PHQ-9) where available. | 1 year
  PHQ-9 scores from 0 to 27, where 1-4 indicates minimal depression and 20-27 indicates severe depression.
Compare changes in sNfL levels with Multiple Sclerosis Quality of Life - 54 (MSQOL-54) physical health summary score where available. | 1 year
  MSQOL-54 scale scores range from 0 to 100 and a higher scale score indicates improved quality of life.
Compare changes in sNfL levels with Multiple Sclerosis Quality of Life - 54 (MSQOL-54) mental health summary score where available. | 1 year
  MSQOL-54 scale scores range from 0 to 100 and a higher scale score indicates improved quality of life.
Compare changes in sNfL levels with magnetic resonance imaging disease activity where available. | 1 year
Compare changes in sNfL levels with changes to multiple sclerosis disease-modifying therapy where available. | 1 year
Correlate changes in sNfL levels with Expanded Disability Status Scale (EDSS) where available. | 1 year
Correlate changes in sNfL levels with Symbol Digit Modalities Test (SDMT) where available. | 1 year
  SDMT scale is from 0 to 110, where 0 indicates none correct and 110 indicates all correct.
Correlate changes in sNfL levels with Patient Health Questionnaire-9 (PHQ-9) where available. | 1 year
  PHQ-9 scores from 0 to 27, where 1-4 indicates minimal depression and 20-27 indicates severe depression.
Correlate changes in sNfL levels with Multiple Sclerosis Quality of Life - 54 (MSQOL-54) physical health summary score where available. | 1 year
  MSQOL-54 scale scores range from 0 to 100 and a higher scale score indicates improved quality of life.
Correlate changes in sNfL levels with Multiple Sclerosis Quality of Life - 54 (MSQOL-54) mental health summary score where available. | 1 year
  MSQOL-54 scale scores range from 0 to 100 and a higher scale score indicates improved quality of life.
Correlate changes in sNfL levels with magnetic resonance imaging disease activity where available. | 1 year
Correlate changes in sNfL levels with changes to multiple sclerosis disease-modifying therapy where available. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Dent Neurologic Institute, Amherst, New York, United States

IPD SHARING:
Plan to Share IPD: No